CLINICAL TRIAL: NCT07370428
Title: Evaluation of the Effectiveness of Ultrasound-Guided Quadro-Iliac Plane Block in Postoperative Analgesia Management Following Lumbar Instrumentation Surgery
Brief Title: US-Guided Quadro-Iliac Plane Block for Postoperative Analgesia After Lumbar Instrumentation
Acronym: QIPB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Merih Yıldız Eglen, Principal Investigator, MD, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BursaCityHOS 1
Record Dates: First submitted 2025-12-26; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain
Keywords: Quadro-Iliac Plane Block; Lumbar Instrumentation Surgery; Pain Management
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group QIPB (Active Comparator): Participants in this arm will receive an ultrasound-guided Quadro-Iliac Plane Block. The block will be performed at the end of surgery, before extubation, with the patient in the prone position under standard sterilization conditions. A convex ultrasound probe will be placed at the level where the quadratus lumborum muscle (QLM) attaches to the iliac crest to visualize the erector spinae muscle (ESM) and the underlying QLM.
  The block location will be confirmed by injecting 2 mL of isotonic solution at the QLM-iliac crest junction. Subsequently, 20 mL of 0.25% bupivacaine will be injected, and the spread of the local anesthetic between the ESM and QLM will be observed under ultrasound guidance. The block will be performed bilaterally with a total volume of 40 mL.
  Interventions: Procedure: Quadro-Iliac Plane Block
- Group Control (No Intervention)

INTERVENTIONS:
Procedure: Quadro-Iliac Plane Block — Ultrasound-guided regional anesthesia technique performed between the erector spinae muscle and the quadratus lumborum muscle at the iliac crest level.
  Arms: Group QIPB

SUMMARY:
Lumbar instrumentation surgery is associated with significant postoperative pain. This study evaluates the analgesic effectiveness of the ultrasound-guided Quadro-Iliac Plane Block in patients undergoing lumbar instrumentation surgery, aiming to assess the efficacy of this newly developed technique for postoperative pain management.

DETAILED DESCRIPTION:
Lumbar instrumentation surgery is associated with significant postoperative pain, which may reduce patient comfort, delay early mobilization, and increase analgesic requirements. Effective postoperative pain management is essential for enhancing recovery and reducing postoperative morbidity. In this context, regional anesthesia techniques have become an important component of multimodal analgesia strategies.

The Quadro-Iliac Plane Block is a newly described ultrasound-guided regional analgesia technique. This block aims to provide effective analgesia by targeting the relevant branches of the lumbar nerves supplying the surgical area. However, clinical evidence regarding its effectiveness in postoperative analgesia following lumbar instrumentation surgery remains limited.

This study aims to evaluate the postoperative analgesic effectiveness of the ultrasound-guided Quadro-Iliac Plane Block in patients undergoing lumbar instrumentation surgery. The findings of this study are expected to contribute to the assessment of this newly developed technique as a safe and effective option for postoperative pain management in lumbar spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Classified as American Society of Anesthesiologists (ASA) physical status I-III
* Scheduled for elective lumbar instrumentation surgery
* Surgery performed under general anesthesia
* Provision of written informed consent

Exclusion Criteria:

* Use of anticoagulant or antiplatelet medications
* Presence of bleeding diathesis or coagulation disorders
* Known allergy or hypersensitivity to local anesthetics or opioid medications
* Infection at the planned block site
* Alcohol or drug dependence
* Cognitive impairment preventing reliable pain assessment using the NRS
* Pregnancy or lactation
* History of previous lumbar spine surgery
* Diabetes mellitus
* Renal or hepatic impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative 48-Hour PCA Opioid Consumption | Postoperative 0-8, 8-16, 16-24, 24-48 intervals
  Total amount of opioid delivered by the patient-controlled analgesia (PCA) device during the first 48 hours after surgery, recorded in milligrams (mg).
QoR-15 Recovery Score | Postoperative 24th and 48th hours
  The investigators will use the Turkish version of Quality of Recovery (QoR) / QoR-15 questionairre
  PART A How have you been feeling in the last 24 hours? (0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent])
  Able to breathe easily Been able to enjoy food Feeling rested Have had a good sleep Able to look after personal toilet and hygiene unaided Able to communicate with Getting support from hospital doctors and nurses Able to return to work or usual home activities Feeling comfortable and in control Having a feeling of general well-being
  PART B Have you had any of the following in the last 24 hours? (10 to 0, where: 10 = none of the time [excellent] and 0 = all of the time [poor]) Moderate pain Severe pain Nausea or vomiting Feeling worried or anxious Feeling sad or depressed

SECONDARY OUTCOMES:
Dynamic and static NRS scores | 0, 2, 4, 8, 16, 24, and 48 hours postoperatively
  Numeric Rating Scale (NRS) (0-10) pain scores at rest or movement at predefined postoperative hours
Total rescue analgesic dose | Postoperative 24th and 48th hours
  Despite the use of patient-controlled analgesia (PCA), if the Numeric Rating Scale (NRS) score is ≥4 at any time point, 0.5 mg/kg intravenous meperidine will be administered as rescue analgesia.
  Total amount of meperidin during the first 24 and 48 hours after surgery, recorded in milligrams (mg).
Time of first request for rescue analgesia | Postoperative 48-Hours
  Despite the use of patient-controlled analgesia (PCA), if the Numeric Rating Scale (NRS) score is ≥4 at any time point, 0.5 mg/kg intravenous meperidine will be administered as rescue analgesia.
Length of Hospital Stay | Patients will remain under observation for at least 2 weeks until their postoperative discharge. Follow-up will be completed upon discharge. The length of hospital stay will be recorded (day).
  Length of hospital stay will be defined as the number of days from the end of surgery to hospital discharge.
Block and Opioid-Related Adverse Effects and Complications | Postoperative 48-Hours
  Block- and opioid-related adverse effects and complications, including but not limited to local anesthetic toxicity, hematoma, infection, nerve injury, nausea, vomiting, pruritus, sedation, and respiratory depression, will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Girit M, Akin T, Narayanan M, Alici HA. Ultrasound guided quadro-iliac plane block: another novel fascial plane block. Pain Med. 2024 May 3;25(6):370-373. doi: 10.1093/pm/pnae018. PMID 38459608
- [Background] Turan EI, Sahin AS. Quadro-iliac plane block (QIPB) in lumbar stabilisation surgeries: A case series. Indian J Anaesth. 2025 Feb;69(2):244-245. doi: 10.4103/ija.ija_1077_24. Epub 2025 Jan 29. No abstract available. PMID 40160919
- [Background] Ciftci B, Cetinkal A, Alver S, Ahiskalioglu A. Quadro-iliac plane block for lumbar multi-level instrumentation surgery: far away from the surgical area. Minerva Anestesiol. 2025 Apr;91(4):358-359. doi: 10.23736/S0375-9393.24.18680-4. Epub 2024 Dec 10. No abstract available. PMID 39656149